CLINICAL TRIAL: NCT07343050
Title: Evaluation of Dental Restorations
Brief Title: Evaluation of the Effect of Flowable Composites on Postoperative Sensitivity in Class I Restorations.
Status: Recruiting | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Muhammet Karadaş, Clinical Professor, Recep Tayyip Erdogan University
Other Study IDs: RTEUDHFMKARADAS005
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Dentin Caries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dental restorations — Composite restorations

SUMMARY:
The aim of this study is to evaluate the effect of flowable conventional and bulk-fill composites on postoperative sensitivity in class I cavities over long-term follow-up. The hypothesis to be tested in this study is that the type of composite material will not affect clinical success.

ELIGIBILITY:
Inclusion Criteria:

* good general health
* no heart disease
* no diabetes
* no systemic diseases such as hypertension

Exclusion Criteria:

* Patients with advanced periodontitis and associated postoperative sensitivity,
* Pregnant and breastfeeding women,
* Patients undergoing orthodontic treatment,
* Patients using appliances,
* Patients with direct pulp capping

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The entire study will be conducted at the Restorative Dentistry Department clinic of the Faculty of Dentistry at Recep Tayyip Erdoğan University. Participants who have received routine dental treatment at the university's dental clinic and whose records are kept will be included in the research.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2027-01-16 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
FDI criteria | 2 years
  good, very good, poor

CONTACTS AND LOCATIONS:
Overall Officials: Elanur Yıldızoğlu, Dr, Principal Investigator — Recep Tayyip Erdogan University
Locations (1):
- Muhammet Karadaş, Merkez, Rize Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No